CLINICAL TRIAL: NCT03065868
Title: Effect of H. Pylori Eradication on the Fate of H. Pylori-associated Gastric Polyp (Randomized Controlled Study)
Brief Title: Effect of H. Pylori Eradication on the Fate of H. Pylori-associated Gastric Polyp
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Su Youn Nam, Clinical professor, Kyungpook National University Chilgok Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KNUMC_15-1045
Record Dates: First submitted 2017-02-18; First posted 2017-02-28 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Gastric Polyp; Helicobacter Pylori Infection
Keywords: gastric polyp; Helicobacter pylori eradication
MeSH Terms: conditions — Polyposis, Gastric | interventions — Clarithromycin

STUDY DESIGN:
Intervention Model Description: open labelled randomized controlled trial. randomization : 2015 September
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eradictaion (Experimental): H. pylori eradication group
  Interventions: Drug: H. pylori eradication (Amoxaxillin, Lanston, Clarithromycin)
- non-eradication (No Intervention): H. pylori non-eradication group

INTERVENTIONS:
Drug: H. pylori eradication (Amoxaxillin, Lanston, Clarithromycin) — H. pylori eradication (Triple Therapy) as first line treatment if eradication failure, quadruple therpy will be provided as 2nd line treatment
  Other Names: Triple Therapy
  Arms: eradictaion

SUMMARY:
Evaluation of the effect of H. pylori eradication on regression of H. pylori-related gastric polyp (Ranomized controlled trial)

1. Study design: open labeled RCT
2. Study group H. pylori eradication group (N=17), non-eradication group (N=15)
3. Treatment plan

   1. Baseline EGD

      : 0.3-1cm sized polyp - bx & CLO test (antrum & body)

      ==> if H. pylori positive and eligible patients, randomization
   2. Triple therapy
   3. UBT (4week after eradication)
   4. Follow-up EGD: gross finding, CLO test
4. Evaluation of polyp regression

   1. disappear
   2. regression over 50% (size, number)
   3. no change or increase (size, number)

DETAILED DESCRIPTION:
(A) Study population

1. inclusion HP-realetd polyp polyp size with 0.3cm-1cm 20 yr - 70yr
2. exclusion peptic ulcer, healing stage or acute stage recent use of PPI within 4weeks Liver cirrhosis, renal insufficiency, other serious chronic or acute disease current infection of other bacteria, virus, or fungus cancer, psychologic disease heavy drinker drug abuser pregnant women, Penicillin allergy, digoxin, antifungal, wafarin previosu H. pylori eradication enroll gastric polyp with bleeding or malignant transformation tiny polyp less than 3mm.

(B) Study method

1. Study design: open labeled RCT
2. Study group H. pylori eradication group (N=17), non-eradication group (N=15)
3. Treatment plan

   1. Baseline EGD: 0.3-1cm sized polyp - bx & CLO test (antrum & body) ==> if H. pylori positive and eligible patients, randomization
   2. Triple therapy
   3. UBT (4week after eradication) if eradication failure in triple therapy, 2nd line treatment (metroniazole based quadraple therpay) and the UBT (4week after eradication)
   4. Follow-up EGD (3-9M): gross finding, CLO test
4. Evaluation of polyp regression

   1. disappear
   2. regression over 50% (size, number)
   3. no change or increase (size, number)
5. Statistical analysis

   1. Chi-square test to compare polyp regression between treatment & control group.
   2. t-test to compare continuous variables between treatment & control group.
   3. Paired T-test to compare the size between baseline and follow-up EGD.
   4. Regression analysis: univariate & multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

* Gastric polyp with current infection of H. pylori
* Gastric polyp size with 3mm-10mm
* Age of 20 yr - 70yr

Exclusion Criteria:

* Gastric ulcer ir duodenal ulcer (healing stage or acute stage)
* Use of PPI within 4weeks
* Liver cirrhosis, renal insufficiency, other serious chronic or acute disease
* Current infection of other bacteria, virus, or fungus
* Any cancer, psychologic disease
* Heavy drinker
* Drug abuser
* Pregnant women
* Penicillin allergy
* Use of digoxin, antifungal, wafarin
* Previous H. pylori eradication
* Gastric polyp with bleeding or malignant transformation
* Tiny polyp less than 3mm.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-12-09 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Compare regression rate of gastric polyps between H. pylori eradication and non-eradication groups. Regression of gastric polyp: one of below 1) Disappearance of gastric polyp 2) Reduction of polyp size over 50% | up to 24months
  Evaluation of the effect of H. pylori eradication on the regression of H. pylori associated gastric polyp
  Study group
  1. H. pylori eradication
  2. H. pylori non-eradication
  Definition of gastric polyp change:
  1. Disappearance of gastric polyp
  2. Reduction of polyp size over 50%
  3. No change of size or increased size

CONTACTS AND LOCATIONS:
Overall Officials: Su Youn Y Nam, MD, PhD, Principal Investigator — Kyungpook National University Medical Center
Locations (1):
- Su Youn Nam, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nam SY, Lee SW, Jeon SW, Kwon YH, Lee HS. Helicobacter pylori Eradication Regressed Gastric Hyperplastic Polyp: A Randomized Controlled Trial. Dig Dis Sci. 2020 Dec;65(12):3652-3659. doi: 10.1007/s10620-020-06065-0. Epub 2020 Jan 23. PMID 31974914